CLINICAL TRIAL: NCT06060132
Title: Risk Analysis of Cardiotoxic Medication Use Due to Sodium Arsenite Chloride Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yi Han, Associate professor of pharmacy, Qianfoshan Hospital
Other Study IDs: YSS001
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Adverse Reaction; Cardiotoxicity; Evaluation Study
Keywords: arsenious acid; arsenic trioxide; cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Arsenic Trioxide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sodium arsenite chloride injection — Patient use of arsenite sodium chloride injection
  Other Names: arsenic trioxide

SUMMARY:
To study the current status of cardiotoxicity of arsenious acid by analyzing the literature, monitoring data, and real-world applications, and to discuss risk factors and preventive and control measures.

DETAILED DESCRIPTION:
Through the project study, the risk rate of cardiotoxicity caused by arsenious acid will be verified and evaluated, and a typical case analysis will be conducted to assess the risk and benefit ratio of clinical use of arsenious acid injection and to formulate preventive measures, so as to guide the holder of the marketing authorization to carry out in-depth safety studies and to ensure the public's safe use of the drug.

ELIGIBILITY:
Inclusion Criteria:

* the period of consultation (for inpatients, according to the time of admission) is from January 1, 2012 to December 31, 2022
* the patient used arsenite sodium chloride injection

Exclusion Criteria:

* Patients with incomplete clinical information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients using sodium arsenite chloride injection from January 1, 2012 to December 31, 2022 approximately 400 people.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
arrhythmia | through study completion, an average of 1 year
  Electrocardiogram shows arrhythmia with marked QT prolongation
adverse reaction | through study completion, an average of 1 year
  All cardiac-related adverse events in the course of the disease regimen
troponin | through study completion, an average of 1 year
  Troponin values
Echocardiogram LVEF | through study completion, an average of 1 year
  Echocardiogram LVEF values

CONTACTS AND LOCATIONS:
Overall Officials: Yi Han, doctorate, Principal Investigator — Qianfoshan Hospital
Locations (2):
- China (2):
  - China, Jinan, Shandong
  - First Affiliated Hospital of Shandong First Medical University ( Qianfoshan Hospital of Shandong Province ), Jinan, Shandong